CLINICAL TRIAL: NCT02718950
Title: Influence of Liraglutide, a GLP-1 Receptor Agonist, on Brown Adipose Tissue (BAT) Activity in Humans
Acronym: i-LAB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Bruno Geloneze, MD, PhD, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i-LAB; U1111-1178-4180 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Brown Adipose Tissue; Hypothalamic Activation; Non-shivering Thermogenesis; Basal Metabolic Rate; Liraglutide; Victoza; Body Composition; Body weight; Adipose Tissue Biopsy
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Body Weight | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liraglutide 3.0 mg (Experimental): Subjects will use liraglutide 3.0 mg for 2 weeks.
  Interventions: Drug: Liraglutide 3.0 mg

INTERVENTIONS:
Drug: Liraglutide 3.0 mg — Subjects will use liraglutide 3.0 mg for 2 weeks
  Other Names: Victoza

SUMMARY:
The purpose of this study is to access liraglutide influence brown adipose tissue recruitment and its thermogenic effect through hypothalamic activation in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index over 30 kg/m2.

Exclusion Criteria:

* Hypersensitivity to liraglutide or any of its vehicle components;
* History of diabetes or pre-diabetes - either by fasting glycemia, oGTT or HbA1c;
* Previous treatment within the last 3 months with glucagon like peptide-1 agonists, iDPP4 or any medication that is associated with BAT activation, including propranolol and benzodiazepines;
* Liver diseases, except non-alcoholic steatohepatitis (NASH);
* Infection by HIV, hepatitis B or hepatitis C;
* Addiction to cannabis, heroin, morphine, cocaine, benzodiazepines or amphetamine;
* Obesity induced by other disorders such as Cushing syndrome, hypothyroidism, lipodystrophy
* Current or history of treatment with medications that may cause significant weight gain within 3 months prior to screening, including systemic corticosteroids (except for a short course of treatment, i.e. 7-10 days), tricyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g. imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium);
* Current participation (or within the last 3 months) in an organized weight reduction program
* Currently or previous using within 3 months before screening of pramlintide, sibutramine, orlistat, topiramate, or metformin (either by prescription or as part of a clinical trial)
* Participation in a clinical trial within the last 3 months prior to screening
* Simultaneous participation in any other clinical trial of an investigational drug
* Previous surgical treatment of obesity;
* Cancer (past or present, except basal cell skin cancer or squamous cell skin cancer), which in the investigator's opinion could interfere with the results of the trial
* Liver enzyme (ALT and AST) above 2.5 x of reference range
* Pancreatic enzymes (amylase, lipase) above 3 x the reference range
* Chronic kidney disease stages 3, 4, or 5
* Relevant inflammatory or acute or chronic infectious disease; hyperthyroidism; neurological, psychiatric, gastrointestinal, respiratory, renal, hepatic or cardiac relevant disease, that could interfere with trial results per the judgment of investigator
* Any condition that at the discretion of investigator could interfere with treatment adhesion on patient safety
* Blood donation or transfusion within the last 3 months
* Pregnancy or intention of pregnancy
* History of Multiple Endocrine Neoplasia Syndrome Type 2 (MEN 2)
* History of pancreatitis
* Less than 80% of liraglutide adherence
* Calcitonin above the reference range at the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of liraglutide administration on brown adipose tissue (BAT) activation in humans | 2 weeks
  Activation of BAT, as considered Standard Uptake Value (SUV) threshold of 2.0 on 18-FDG-PET CT, prior to liraglutide use and after 2 weeks on liraglutide 3.0 mg

SECONDARY OUTCOMES:
Evaluate the effect of liraglutide administration on hypothalamic activation in humans | 2 weeks
  Evaluate the effect of liraglutide administration on hypothalamic tract activation as assessed by magnetic resonance image in humans prior and after 2 weeks on liraglutide 3.0 mg
Evaluate the effect of liraglutide administration on non-shivering thermogenesis in humans | 2 weeks
  Evaluate the effect of liraglutide administration on non-shivering thermogenesis by infrared thermography and indirect calorimetry in humans prior and after 2 weeks on liraglutide 3.0 mg
Evaluate the effect of liraglutide administration on body weight in humans | 2 weeks
  Evaluate the effect of liraglutide administration on total body weight (kg) in humans prior and after 2 weeks on liraglutide 3.0 mg
Evaluate the effect of liraglutide administration on metabolic basal rate in humans | 2 weeks
  Evaluate the effect of liraglutide administration on basal kilocalories/day in humans prior and after 2 weeks on liraglutide 3.0 mg
Evaluate the effect of liraglutide administration on body composition in humans | 2 weeks
  Evaluate the effect of liraglutide administration on lean mass and fat percentage as assessed by dual x-ray absorptiometry (DXA) in humans prior and after 2 weeks on liraglutide 3.0 mg

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, MD, PhD, Principal Investigator — University of Campinas; Lício A Velloso, MD, PhD, Principal Investigator — University of Campinas; José C Lima Júnior, MD, Study Chair — University of Campinas; Riobaldo M Cintra, MD, Study Chair — University of Campinas

IPD SHARING:
Plan to Share IPD: No